CLINICAL TRIAL: NCT01377831
Title: An Open Label, Two Way Crossover Study to Evaluate the Bioavailability and Clinical Tolerability of a Novel Sublingual Wafer Formulation of Ketamine in Healthy Male Volunteers
Brief Title: Study of Ketamine Administered Intravenously and by Sublingual Wafer
Status: Completed | Type: Observational
Sponsor: iX Biopharma Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: KET001
Record Dates: First submitted 2011-06-19; First posted 2011-06-21 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be drawn into Vacuette brand, lithium heparin separator tubes (green/yellow top).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To determine the rate and extent of of absorption of racemic ketamine from sublingual wafer

DETAILED DESCRIPTION:
1. To determine the apparent rate of disintegration of the sublingual wafer
2. To determine the overall clinical tolerability of ketamine when administered as a single dose via the sublingual route. Tolerability will be assessed using a range of objective and subjective parameters as assessed using modified Likert and Bond and Lader scales.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males aged 18-65 years.
2. Good general health without clinically significant renal, hepatic, cardiac or respiratory disease, as determined by the Principal Investigator.
3. Good general mental health as determined by scores on the Symptom Checklist-90-R (SCL-90-R®), a screening instrument which evaluates a broad range of psychological problems and symptoms of psychopathology.
4. Agree to and be capable of signing an Informed Consent Form.
5. Have suitable venous access for blood sampling.
6. BMI within the range of 19-30 kg/m2.

Exclusion Criteria:

1. Renal impairment as evidenced by estimated creatinine clearance (CrCl), measured by the Cockcroft-Gault method, of less than 90 mL/min.
2. Have a laboratory value at the Screening Visit that is outside the normal range, unless it is judged by the Investigator as not clinically significant after appropriate evaluation.
3. A score of more than two standard deviations from the mean on any of the key nine scales in the SCL-90-R ®
4. Any medical condition that in the opinion of the Investigator may adversely impact on the participant's ability to complete the study, including but not limited to:

   * History of cerebral trauma or stroke
   * History of seizure or epilepsy
   * Hyperthyroidism
   * Recent clinically significant URTI (within two weeks of Day 1) or respiratory infection
   * History of Myocardial Infarction or clinically significant cardiac disease including cardiac arrhythmia.
   * Poorly controlled hypertension - as assessed by the Principal Investigator.
   * Clinically significant history of asthma requiring regular supportive or preventative therapy (childhood asthma that has resolved >5 years previously may be suitable for inclusion at the discretion of the Investigator.
   * Glaucoma
5. Plasma AST, ALT and ALP tests in excess of 1.5 times the upper limit of normal.
6. History of severe allergic or anaphylactic drug-related reactions.
7. History of hypersensitivity to ketamine or any of its excipients.
8. Current (within the last six months) clinically significant psychiatric disorder including anxiety, psychosis or depression.
9. Concurrent use of other medication on a regular or daily basis including but not limited to, theophylline, benzodiazepines, thyroxine, sedatives or anti-anxiolytics.
10. Participation in another clinical trial of an investigational agent within 30 days of study entry.
11. Known history of past or present infection with hepatitis C virus (HCV), hepatitis B or human immunodeficiency virus (HIV).
12. Clinically significant abnormal ECG (12-lead) at the screening visit or prior to dosing on Day 1, as determined by the Investigator.
13. Participants who have a marked prolongation of the QT corrected (QTc) interval (i.e., repeated demonstration of a QTc >430 msec for males) at screening or prior to dosing on Day 1 in either study period will not be allowed to continue in the study.
14. Significant history of illicit drug or alcohol use or abuse (as determined by the Principal Investigator).
15. Any alcohol use within 24 hours prior to dosing on Day 1 in each of the study periods.
16. Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the participant returning for follow-up visits on schedule.
17. Blood donation (1 unit or more) within 1 month prior to the screening visit.
18. Current or previous tobacco user (within 12 months prior to Day 1) .
19. Planned surgical procedure requiring general anaesthesia during the study period and within two weeks of study completion

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 8 Healthy Male Volunteers
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Bioavailability of a single 25 mg dose of sublingual (SL) ketamine | 24 hours post-dose for two dosing periods, which were separated by 7 days.
  Bioavailability determined by evaluation and comparison of PK variables following SL and IV administration.

SECONDARY OUTCOMES:
General clinical tolerability and safety | 24 hours post-dose for two dosing periods, which were separated by 7 days.
  Determined by using a range of objective and subjective parameters.
Rate of disintegration | 5 minutes post-dose
  Measured the apparent rate of disintegration of a single 25 mg sublingual wafer formulation of ketamine.

CONTACTS AND LOCATIONS:
Overall Officials: Pual Rolan, Principal Investigator — Pain and Anaesthesia Research Clinic - PARC
Locations (1):
- Pain and Anaesthesia Research Clinic (PARC), Royal Adelaide Hospital, Adelaide, South Australia, Australia